CLINICAL TRIAL: NCT01735539
Title: Dysfunction of Nutritive Blood Flow as a Determinant of Anabolic Resistance in Older People; The Role of Essential Amino Acids in Modulating Muscle Protein Metabolism; Bolus vs. Pulse Feeding Strategies and the Ability of Arginine to Rejuvenate Microvascular Responsiveness.
Brief Title: Dysfunction of Nutritive Blood Flow as a Determinant of Anabolic Resistance With Age; the Role of Amino Acids in Modulating Muscle Metabolism
Acronym: Ajinomoto1A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNottingham F/3/2009
Record Dates: First submitted 2012-11-22; First posted 2012-11-28 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Old Age (Focus; Not a Recognized Condition)
Keywords: old age; sarcopenia; essential amino acid; arginine; contrast enhanced ultrasound; muscle microcirculation; muscle protein synthesis
MeSH Terms: conditions — Sarcopenia | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Old Bolus (Experimental): 15g EAA bolus
  Interventions: Dietary Supplement: 15g EAA bolus
- Old Arginine (Experimental): 15g EAA Bolus supplemented with 3g Arginine
  Interventions: Dietary Supplement: 15g EAA Bolus supplemented with 3g Arginine
- Young Bolus (Experimental): 15g EAA bolus
  Interventions: Dietary Supplement: 15g EAA bolus
- Young Pulse (Experimental): 4 x 3.75g Mixed EAA Pulses
  Interventions: Dietary Supplement: 4 x 3.75g Mixed EAA Pulses
- Old Pulse (Experimental): 4 x 3.75g Mixed EAA Pulses
  Interventions: Dietary Supplement: 4 x 3.75g Mixed EAA Pulses

INTERVENTIONS:
Dietary Supplement: 15g EAA bolus — Oral; in aqueous solution
  Other Names: Mixed Essential Amino Acids
  Arms: Old Bolus; Young Bolus
Dietary Supplement: 4 x 3.75g Mixed EAA Pulses — Oral; in aqueous solution
  Arms: Old Pulse; Young Pulse
Dietary Supplement: 15g EAA Bolus supplemented with 3g Arginine — Oral; in aqueous solution
  Arms: Old Arginine

SUMMARY:
The investigators plan to measure changes in muscle protein metabolism in response to feeding, comparing between a single large essential amino acid (EAA) feed (the normal building blocks of protein) and the provision of the same dose in 4 smaller feeds at 45min intervals. The investigators will perform this study in healthy older (65-75y) and younger (18-28) men. The investigators will also explore how feeding affects muscle blood flow as this is important in the delivery of the nutrients we eat to the muscle where they are used.

The investigators plan to supplement the feed with arginine, a safe and widely found non-essential amino acid, to explore if this can improve muscle blood flow.

DETAILED DESCRIPTION:
We will provide a 15g mixed essential amino acid feed or 4 x 3.75g.

There is sexual dimorphism thus initially we will just recruit males. Powering calculations dictate n=8 in each group.

We will use well established stable isotope tracer techniques (with 13C6 Phenylalanine) to measure muscle protein synthesis and breakdown by Gas Chromatography - combustion - isotope ratio mass spectroscopy.

We will measure leg blood flow by phase shift Doppler and muscle microvascular flow by contrast enhanced ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* age 65-75 or 18-28

Exclusion Criteria:

* BMI >30
* Diabetes
* Beta blocker or steroid use
* Established cerebrovascular, peripheral vascular or ischaemic heart disease.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Muscle Protein Synthesis (FSR, fractional synthetic rate, %/hr) | Across 6hr study
  We measure FSR when fasted and again 0-90, 90-180 and 180-240 post feed.

SECONDARY OUTCOMES:
Muscle Protein Breakdown (MPB) | Across 6hr study
  MBP is measured during fasting and 0-90, 90-180 and 180-240mins post feed.
Whole leg blood flow | Across a 6hr study
  We measure common femoral blood flow by doppler ultrasound when fasted and again 0-90, 90-180 and 180-240 post feed.
Muscle Microvascular Blood flow | Across a 6hr study
  We measure muscle microvascular flow using contrast enhanced ultrasound when fasted and again 0-90, 90-180 and 180-240 post feed.

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Atherton, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham School of Graduate Entry Medicine and Health, Derby, United Kingdom

REFERENCES:
- [Derived] Mitchell WK, Phillips BE, Williams JP, Rankin D, Lund JN, Smith K, Atherton PJ. A dose- rather than delivery profile-dependent mechanism regulates the "muscle-full" effect in response to oral essential amino acid intake in young men. J Nutr. 2015 Feb;145(2):207-14. doi: 10.3945/jn.114.199604. Epub 2014 Dec 10. PMID 25644339